CLINICAL TRIAL: NCT06255925
Title: A Strength-Based Employment Maintenance Program for Individuals on the Autism Spectrum
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: E-1199-22
Record Dates: First submitted 2024-01-16; First posted 2024-02-13 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Autism
Keywords: Autism, Autism Spectrum Disorder, ASD
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder | interventions — Gene Expression

STUDY DESIGN:
Intervention Model Description: Kessler Foundation Strength Identification and Expression (KF-STRIDE® Into Work!)
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): In this arm, participants would participate in in an intervention program that uses character strengths to improve job maintenance skills in young adults.
  Interventions: Behavioral: KF-STRIDE® Into Work!
- Control Group (No Intervention): In this arm, participants are services as usual and will participate in their regular activities.

INTERVENTIONS:
Behavioral: KF-STRIDE® Into Work! — Treatment group will receive 10 web based sessions of a strength-based training tool(once or twice a week). Sessions are approximately 60 minutes long.
  Other Names: Kessler Foundation Strength Identification and Expression
  Arms: Treatment Group

SUMMARY:
The investigators are looking to evaluate how effective a training program that focuses on character strengths may be in improving job maintenance skills in young adults. The investigators are examining the effects of this intervention in young adults who feel they would like to help in improving their satisfaction with work, and in keeping their jobs.

DETAILED DESCRIPTION:
Individuals with autism possess employable and valuable strengths and abilities. Unfortunately, despite these strengths, individuals with autism experience challenges in obtaining and maintaining employment. Traditionally, the majority of interventions designed for autism (including those focused on employment) focus on remediating deficits, without harnessing the strengths of those with autism. This deficit-based approach (i.e. to fix what is deficient in a person with autism) has triggered increasing criticism and dissatisfaction from the autism community. A growing shift toward strength-based training tools represent a holistic approach to treatment of autistic individuals by acknowledging and using their strengths to improve outcomes. To date, no strength-based employment programs have been examined in individuals with autism. Thus, in the current project, the investigators aim to develop and test a strength-based employment program. At Kessler Foundation, the investigators have developed a strength-based training tool: Kessler Foundation Strength Identification and Expression (KF-STRIDE®) which targets job interview skills by teaching individuals with autism to identify and express their personal strengths to a future employer. In the current proposal, the investigators aim to adapt this program to specifically target job maintenance skills.

ELIGIBILITY:
Inclusion Criteria:

* Lives in the United States of America
* Between the ages of 14-26
* Speaks English well and at a 4th grade reading level

Exclusion Criteria:

* Had a stroke, Traumatic Brain Injury, or neurological injury or disease in the past(like brain tumor or epilepsy)
* Has a history of significant psychiatric illness(like schizophrenia or psychosis)
* Has uncontrolled seizures or other unstable medical complications

Ages: 14 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Parent Report Employment Questionnaire | Baseline, Immediate Post-test between weeks 7 and 8
  Consists of questions answered by parents regarding employment difficulties in their children . Questions of employment valued by yes or no, with yes being valued higher. And amount of hours worked from 0-40, with higher score indicating a better outcome.
Work Self-Efficacy Scale | Baseline, Immediate Post-test between weeks 7 and 8
  10 items, scores range from 10-50 with higher scores indicating perceived work capability.
Strengths Self-Efficacy Scale | Baseline, Immediate Post-test between weeks 7 and 8
  Measures the level of one's confidence in her/his ability to practice and apply her/his strengths. 34 items, scores range from 0-340
Strengths Knowledge and Strengths Use Scale(SKUS) | Baseline, Immediate Post-test between weeks 7 and 8
  Measure to assess knowledge and use of one's strengths and measure changes following strengths-based interventions. Two scores: Strengths Use and Strengths Knowledge. Strengths Use values range from 14-98, with higher score indicating a better outcome. Strengths Knowledge values range from 8-56, with higher score indicating a better outcome.
Flourishing(FS) | Baseline, Immediate Post-test between weeks 7 and 8
  Measure of well-being and "flourishing". Values range from 8-56, with higher score indicating a better outcome.
Patients Global Impression of Change | Baseline, Immediate Post-test between weeks 7 and 8
  Measure of perception of intervention resulting in meaningful change for a participant's life. 6 Items, with higher score indicating effectiveness of positive change.
Intervention Effectiveness From Participant Point | Baseline, Immediate Post-test between weeks 7 and 8
  Measure of perception of intervention resulting in meaningful change for a participant's life. 15 Items, with higher score indicating effectiveness of positive change.

SECONDARY OUTCOMES:
Minnesota Work Satisfaction | Baseline, Immediate Post-test between weeks 7 and 8
  20 item part 1, scores range from 20-100. Measure of present job satisfaction, with higher scores indicating higher job satisfaction. 8 item part 2 with open-ended questions, there is no maximum or minimum.
Job search | Baseline, Immediate Post-test between weeks 7 and 8
  12 item, 0-60 with the higher score indicating the greater level of job search behaviors.
Search for Work Self-Efficacy Scale | Baseline, Immediate Post-test between weeks 7 and 8
  12 items, scores range from 12-60. Items concern one's perception of their capability to select among job offers, to build strategies for the attainment of a goal, to respect other people's competences, and to work with new members, to manage time difficulties, and stressful situations typical of job searches, to consider a failure a challenge rather than a problem.
Connor- Davidson Resilience Scale(CD-RISC) | Baseline, Immediate Post-test between weeks 7 and 8
  10 items, scores range from 0 to 40. Lower scores indicate less resilience and higher scores indicate greater resilience.
Voicemail Elicitation Task(VET)/ Email Elicitation Task(EET) | Baseline, Immediate Post-test between weeks 7 and 8
  Measures how individuals respond to social situations using politeness/impoliteness. Values are calculated by dividing the total number of politeness markers by the total time in minutes, with a higher score indicating a better outcome. There are no minimum or maximum values for this test.
Work Chat Assessment | Baseline, Immediate Post-test between weeks 7 and 8
  Measure of work place appropriate behavior. Participants interact with a virtual human avatar in various scenarios. Higher scores indicate more appropriate work place behavior. Minimum of 0 and Maximum of 100.
Rosenberg Self-Esteem Scale(RSES) | Baseline, Immediate Post-test between weeks 7 and 8
  Self-report self-esteem questionnaire. Values range from 10-40, with higher score indicating better outcome.
Twenty Statements Task | Baseline, Immediate Post-test between weeks 7 and 8
  20-item questionnaire used to measure an individual's self concept filling out the twenty items that each start with the words "I am..." which will be analyzed for positive and negative valence, with higher score indicating a better outcome. There is no maximum or minimum value for this test.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Genova, Ph. D., Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No